CLINICAL TRIAL: NCT05729698
Title: Efficacy of A Novel in Prevention of Neonatal Hypothermia in Preterm: Baby Warmer Swaddle
Brief Title: Efficacy of A Novel in Prevention of Neonatal Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Caglar, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sedacaglar
Record Dates: First submitted 2023-01-16; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Hypothermia; Newborn; Preterm Birth
Keywords: hypothermia; newborn; body temperature changes; preterm birth
MeSH Terms: conditions — Hypothermia; Premature Birth; Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polyethylene bag method (Experimental): polyethylene bag method: preterm babies will be placed in polythene bags after birth
  Interventions: Other: polyethylene bag
- baby warmer swaddle method (Experimental): baby warmer swaddle group: preterm babies will be placed in baby warmer swaddle after birth
  Interventions: Device: Baby warmer swaddle

INTERVENTIONS:
Device: Baby warmer swaddle — Baby Swaddle with Heating System
  Other Names: prethermo
  Arms: baby warmer swaddle method
Other: polyethylene bag — polyethylene food bag
  Arms: polyethylene bag method

SUMMARY:
The research was carried out to determine the effect of baby warmer swaddle, which has a heating system used after the birth of preterm babies, on the development of hypothermia.

Design: Randomized controlled clinical trial Setting: The research was carried out in the NICU of a training and research hospital in Istanbul.

Method: A total of 65 babies between 32-37 weeks of gestation were included in the study. In accordance with the routine procedure of the clinic, preterm babies wrapped in polyethylene bags after birth formed the control group (n=33), while babies wrapped in polyethylene bags and placed in a swaddle with a heating system formed the experimental group (n=32).

DETAILED DESCRIPTION:
Although neonatal hypothermia has higher rates especially in underdeveloped and developing countries, it is a global health problem also seen in developed countries. In a meta-analysis study, the prevalence of neonatal hypothermia was reported as 57.2% in East Africa. In a multicenter, prospective study, 79.6% of preterm newborns were admitted to NICUs with hypothermia in Ethiopia. In a study, the incidence of hypothermia to be 53% in the first 24 hours of life in preterm infants they conducted in a hospital in France. In a study, in 28 countries with upper-middle income status, admission temperature data of a total of 454,617 very low birth weight infants from 2009 to 2016 were analyzed. Although these data showed an improvement in hypothermia rates ranging from 52.6% (2009) to 38.2% (2016), approximately 4 out of 10 infants experienced hypothermia when admitted to the NICU. Similarly, in the United Kingdom, the National Neonatal Monitoring Program reported the prevalence of hypothermia as 28% and 25% for babies born in 2015 and 2016, respectively, emphasizing hypothermia as an ongoing problem.

ELIGIBILITY:
Inclusion Criteria: Preterms;

* between 32-37 GH,
* with an indication for hospitalization in the NICU,
* with a body temperature of 36.4 °C and above in the axillary route immediately after birth,
* with a maternal body temperature between 36.4 °C and 38 °C in the tympanic route are included in the study

Exclusion Criteria: preterms;

* with congenital anomalies,
* who were transported to another hospital, or who were transported to the hospital where the research was conducted from an external center

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Neonatal hypothermia | immediately after birth
  Neonatal hypothermia is defined as temperature < 36.5C
Neonatal hypothermia | 20 minutes after birth
  Neonatal hypothermia is defined as temperature < 36.5C
Neonatal hypothermia | 40 minutes after birth
  Neonatal hypothermia is defined as temperature < 36.5C
Neonatal hypothermia | 60 minutes after birth
  Neonatal hypothermia is defined as temperature < 36.5C

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No